CLINICAL TRIAL: NCT05928338
Title: Feasibility of a Peer-Supported, WhatsApp-Assisted, Lifestyle Modification Intervention for Weight Reduction Among Adults in an Urban Slum of Karachi, Pakistan: A Mixed-Methods, Single Group, Pretest-Posttest, Quasi-Experimental Study
Brief Title: Lifestyle Modification for Weight Reduction With Peer Support Among Adults in an Urban Slum of Karachi, Pakistan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Romaina Iqbal, Associate Professor and Section Head Non-Communicable Diseases and Mental Health, Aga Khan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-3550-9021
Record Dates: First submitted 2023-06-14; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Weight Loss
Keywords: Lifestyle modification; Peer support; Weight reduction; Slums; WhatsApp; Mixed-methods
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peer-supported, WhatsApp assisted lifestyle modification intervention (Experimental): Study participants with BMI 23 kg/m2 and above was provided with a lifestyle modification intervention supported by peers for modifying their diet and increase physical activity to reduce weight
  Interventions: Behavioral: Peer-supported, WhatsApp-assisted lifestyle modification intervention

INTERVENTIONS:
Behavioral: Peer-supported, WhatsApp-assisted lifestyle modification intervention — The lifestyle modification intervention, supported by peers and WhatsApp voice calls aimed to assist participants in making dietary modifications, increasing physical activity, and achieve a weight loss of 5% of their initial body weight as well as avoid weight gain. A trained nutritionist delivered the intervention after the baseline assessment individually or in groups that covered six sessions related to dietary modifications, physical activity, set-up goals and action plans, and peer assignments and then once monthly for a year using WhatsApp voice calls to the participants and peers.

SUMMARY:
The feasibility study was conducted using a mixed-methods single group, pre and post-test design (Quasi experiment) approach. The investigator assessed if a weight reduction program using WhatsApp and peer support would work well enough to conduct a larger study. The investigator conducted the study in an urban slum (Azam Basti) in Karachi, Pakistan and enrolled 50 participants, along with participant nominated peers from the same family. Initial eligibility was assessed over the phone. Those who met the initial eligibility were visited to assess eligibility in terms of BMI (23 kg/m2 and above). Height was measured in centimeters (cm) and weight in kilograms (kgs) using a digital weighing scale. Both values were entered into the web-based calculator to calculate BMI. Participants with a BMI of 23 kg/m2 and above were enrolled and written informed consent was obtained. The participants then nominated one peer from the family. Peer eligibility was assessed and written informed consent was obtained. Once the participants and peers were enrolled in the study, the baseline assessments were completed. During the baseline assessments, participants were interviewed for sociodemographic and health-related information, 24-hour dietary recall, and Global Physical Activity Questionnaire (GPAQ). Peers were also interviewed for sociodemographic information. After the baseline assessment, the participants and peers received lifestyle modification education through WhatsApp voice calls for three days and then once monthly for one year delivered by a trained nutritionist. The intervention was delivered mostly in groups. The peer-supported lifestyle modification intervention was developed with the aim of helping participants adopt healthier lifestyles by making dietary changes, increasing physical activity, and achieving a weight loss goal of 5% of their initial body weight. Additionally, the intervention aimed to prevent weight gain among participants. The participants were followed-up for one year. Participants weight (kg), diet through 24-hour dietary recall, and physical activity through Global Physical Activity Questionnaire (GPAQ) were assessed every month. Social support questionnaire was also asked from participants at 3, 6, 9, and 12 months. The investigator also conducted in-depth interviews at the end of the study with study participants and peers to understand the barriers, facilitators, and experiences of the lifestyle modification intervention program.

ELIGIBILITY:
Inclusion Criteria for Participants:

* Males and females
* Aged 20 to 60 years
* Had access to smartphones and an internet connection
* Agreed to nominate one peer from their family
* Provide written informed consent

Exclusion Criteria for Participants:

* Pregnancy
* Chronic conditions, disability, and other health-related issues that require special treatment and dietary and physical activity restrictions

Eligibility Criteria for Peers:

* Males and females
* Aged 20 years and above
* Willing to attend online training sessions
* Agreed to help participants with lifestyle modification adherence throughout the study
* Provide written informed consent

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Number of participants screened, recruited, retained, and responded to monthly interviews | one year
  The feasibility of the study was evaluated by reporting number of participants screened, recruited, retained, and responded to monthly interviews
Barriers, facilitators, acceptability, and experience of participants and peers to lifestyle modification intervention through in-depth interviews | one year
  In-depth interviews were conducted at the end of the study to explore barriers, facilitators, acceptability, and experience of participants and peers about lifestyle modification intervention for weight reduction
Change in mean weight in kilograms | one year
  Trends of change in mean weight in kilograms was evaluated throughout the study
Change in mean calorie intake (kcal/day) from food using 24-hour dietary recall | one year
  Trends of change in mean calorie intake (kcal/day) from food using 24-hour dietary recall was evaluated throughout the study
Change in mean calorie expenditure (kcal/day) through physical activity using Global Physical Activity questionnaire (GPAQ) | one year
  Trends of change in mean calorie expenditure (kcal/day) through physical activity using Global Physical Activity questionnaire (GPAQ) was evaluated throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Romaina Iqbal, Ph.D, Principal Investigator — Aga Khan University
Locations (1):
- Sabahat Naz, Karachi, Pakistan

REFERENCES:
- [Derived] Naz S, Haider KA, Jaffar A, Khan U, Azam I, Siddiqui AR, Iqbal R. Feasibility of a peer-supported, WhatsApp-assisted, lifestyle modification intervention for weight reduction among adults in an urban slum of Karachi, Pakistan: a mixed-methods, single-group, pretest-post-test, quasi-experimental study. BMJ Open. 2023 Aug 1;13(8):e070913. doi: 10.1136/bmjopen-2022-070913. PMID 37527890